CLINICAL TRIAL: NCT00063960
Title: A Phase II Trial Of Toxicity Assessment In Two Cohorts Of Patients (Resection Alone Or Ablation With Or Without Resection Of Hepatic Metastases From Colorectal Cancer) Treated With Adjuvant Hepatic Arterial Infusion (HAI) FUDR Plus Systemic CPT-11
Brief Title: Hepatic Arterial Infusion With Floxuridine and Systemic Irinotecan After Surgery in Treating Patients With Hepatic (Liver) Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z05032; ACOSOG-Z05032; CDR0000305857 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; stage IV rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Floxuridine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- floxuridine + irinotecan (Experimental): Within 4-8 weeks after prior resection or ablation, patients receive hepatic arterial infusion of floxuridine continuously on days 1-14 and irinotecan IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of unacceptable toxicity.
  Patients are followed every 3 months for 2 years.
  Interventions: Drug: floxuridine; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: floxuridine
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as floxuridine and irinotecan use different ways to stop tumor cells from dividing so they stop growing or die. Hepatic arterial infusion uses a catheter to deliver chemotherapy directly to the liver. Combining more than one drug and giving them in different ways may kill any tumor cells remaining after surgery.

PURPOSE: Phase II trial to study the effectiveness of systemic irinotecan and hepatic arterial infusion with floxuridine after surgery in treating patients who have hepatic (liver) metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of hepatic arterial infusion with floxuridine and systemic irinotecan adjuvant to liver metastases resection or ablation with or without resection in patients with hepatic metastases secondary to colorectal cancer.
* Determine the overall survival of patients treated with this regimen.
* Determine the time to any hepatic recurrence or progression in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to prior therapy (liver metastases resection only vs ablation with or without resection).

Within 4-8 weeks after prior resection or ablation, patients receive hepatic arterial infusion of floxuridine continuously on days 1-14 and irinotecan IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of unacceptable toxicity.

Patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic colorectal adenocarcinoma

  * Primary colorectal adenocarcinoma that has been completely resected (R0 disease)

    * No evidence of residual, viable tumor by abdominal/pelvic helical CT scan or MRI with IV contrast
  * Metastatic disease

    * No more than 9 liver metastases
    * All lesions completely resected or completely treated by ablation (with or without resection)

      * All lesions treated by ablation must have been less than 5 cm in size and at least 5 mm away from main/left/right portal vein, common bile duct, and inferior vena cava
      * All resected lesions must have a negative surgical margin (R0)
* Disease progression after prior systemic irinotecan for metastatic disease allowed
* No extrahepatic metastases confirmed by chest CT scan except colorectal mesenteric lymph node metastases resected at the time of primary tumor resection

  * No other prior resection of extrahepatic metastases
* Must have the entire liver remnant perfused with a single catheter
* Must have a nuclear medicine macro-aggregated albumin flow scan to confirm the area of pump perfusion before study registration

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2 mg/dL
* Alkaline phosphatase no greater than 2.0 times upper limit of normal (ULN)
* AST and ALT no greater than 2.0 times ULN
* No active hepatitis B or C infection
* No histological evidence of cirrhosis

Renal

* Creatinine no greater than 1.5 times ULN
* Calcium less than 1.3 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

  * Postmenopausal women must be amenorrheic for at least 12 consecutive months to be deemed not fertile
* Medically fit to begin chemotherapy between 4 and 8 weeks after surgery
* Prior cancer allowed if all of the following criteria are met:

  * Undergone potentially curative therapy for all prior malignancies
  * No other malignancy within the past 5 years except the following:

    * Effectively treated basal cell or squamous cell skin cancer
    * Carcinoma in situ of the cervix that has been effectively treated by surgery alone
    * Lobular carcinoma in situ of the ipsilateral or contralateral breast treated by surgery alone
  * No evidence of recurrence of any prior malignancy
* No prior hepatic arterial infusion pump malfunction, malperfusion, or infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunologic or biologic therapy

Chemotherapy

* No prior chemotherapy within 4 weeks before hepatic resection or hepatic ablation (with or without resection)
* No prior hepatic arterial infusion with fluorouracil or floxuridine

Radiotherapy

* No concurrent adjuvant radiotherapy to the pelvis
* No other concurrent radiotherapy

Other

* No other concurrent systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2003-08; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 2 years

SECONDARY OUTCOMES:
time to hepatic recurrence or progression | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuman Fong, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Integris Oncology Services, Oklahoma City, Oklahoma
  - University Medical Group, Providence, Rhode Island